CLINICAL TRIAL: NCT04418817
Title: An Assessment of the Safety and Performance of the Modulus® 3D-printed Titanium Interbody Implant in Patients Undergoing eXtreme Lateral Interbody Fusion (XLIF®)
Brief Title: Modulus in XLIF Study
Status: Completed | Type: Observational
Sponsor: NuVasive (Industry)
Responsible Party: Sponsor
Organization: Globus Medical Inc (Industry)
Other Study IDs: NUVA.X1901
Record Dates: First submitted 2020-06-02; First posted 2020-06-05 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Degenerative Disc Disease; Degenerative Spondylolisthesis; Degenerative Scoliosis
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | US Export: No

GROUPS / COHORTS (1):
- Modulus XLIF Interbody System

SUMMARY:
The primary objective of this study is to evaluate the safety and performance of the Modulus 3D-printed titanium interbody implant in patients undergoing thoracic and/or lumbar XLIF as measured by reported complications, radiographic outcomes, and patient-reported outcomes.

DETAILED DESCRIPTION:
Patients considered for this study will have previously undergone surgery for their spinal condition according to the standard of care of the practitioner. All patients at a given site who meet eligibility requirements will be asked to consent to participate in the study. Once enrolled in the study, subjects will undergo a computed tomography (CT) scan at 12 months postoperative or later to evaluate their fusion status. If the patient already had a postoperative CT scan at 12 months or greater, this will be used in this study and an additional CT scan should not be performed for this study. Available progress notes, medical records, patient-reported outcomes, radiographs (plain film and CT scans, if available), and complications will be obtained from the medical records of all enrolled subjects.

The safety and performance of the Modulus XLIF interbody implant will be assessed using the following:

1. Complications attributable to the use of the Modulus XLIF interbody implant as noted in surgical summaries, progress notes, and hospital records
2. Radiographic outcome (fusion) and description of device status from plain film radiographs and CT scan(s)
3. Neurologic status, symptoms, and/or subject self-reported clinical outcomes (e.g., pain and disability), as available

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients who are ≥18 years of age at the time of surgery
2. Treated with XLIF procedure with the Modulus 3D-printed titanium interbody implant at:

   1. One or two thoracic and/or lumbar levels for degenerative disc disease or degenerative spondylolisthesis, or
   2. Any number of thoracic and/or lumbar levels for degenerative scoliosis (defined as >10º coronal curve)
3. Interbody fusion with autograft and/or allograft
4. Any NuVasive supplemental fixation
5. Patient is able and to undergo a CT scan. If the patient already had a postoperative CT scan at 12 months or greater, this will be used in this study and an additional CT scan should not be performed for this study.
6. Patient understands the conditions of enrollment and is willing to sign an informed consent form to participate.

Exclusion Criteria:

1. Use of any bone graft with the Modulus XLIF interbody implant that is not FDA-cleared for use in the interbody space. Examples of these include:

   1. Bone morphogenetic protein (BMP) (e.g., Infuse (Medtronic))
   2. Synthetic bone graft extenders (e.g., AttraX (NuVasive), Formagraft (NuVasive), Mastergraft (Medtronic), Vitoss (Stryker), Actifuse (Baxter), nanOss (RTI Surgical), Fibergraft (Prosidyan/Depuy Synthes), ChronOs (Depuy Synthes))
   3. Demineralized bone matrices (DBM) regulated as medical devices by the FDA (e.g., Grafton Putty/Gel (Medtronic), DBX (MTF/Depuy Synthes), Accell Evo3 (IsoTis), Propel Putty/Gel (NuVasive))
   4. Peptide enhanced bone graft (e.g., iFactor (Cerapedics))
2. Previous lumbar fusion surgery at the currently treated level(s) (adjacent-level surgery is acceptable)
3. Patients with active infection at the surgical site at the time of surgery
4. Patient is involved in active litigation relating to the spine (worker's compensation claim is allowed if it is not contested)
5. Patient is unwilling or unable to undergo a CT scan due to pregnancy or other medical condition
6. Patient is a prisoner
7. Patient is participating in another clinical study that would confound study data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients considered for this study will have previously undergone surgery for their spinal condition according to the standard of care of the practitioner. All patients at a given site who meet eligibility requirements will be asked to consent to participate in the study. Once enrolled in the study, subjects will undergo a computed tomography (CT) scan at 12 months postoperative or later to evaluate their fusion status.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2020-03-22 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Rate of Complications | At least 12 months
  Rate of complications attributable to use of the Modulus XLIF interbody implant
Proportion of subjects with apparent radiographic fusion at 12 months or greater postoperative | At least 12 months
  Proportion of subjects with fusion at 12 months or greater

SECONDARY OUTCOMES:
Improvement in neurologic status | At least 12 months
  Proportion of subjects with neurological improvement as compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Malone, MS, Study Director — NuVasive
Locations (2):
- United States (2):
  - Erik C. Spayde, MD Inc., Thousand Oaks, California
  - Georgia Spine & Neurosurgery Center, Atlanta, Georgia